CLINICAL TRIAL: NCT03303027
Title: Use of 6-0 Fast Absorbing Gut Versus 5-0 Fast Absorbing Gut for Linear Cutaneous Wound Closure: a Randomized Evaluator Blind Split Wound Comparative Effectiveness Trial.
Brief Title: 6-0 Fast Absorbing Gut Versus 5-0 Fast Absorbing Gut for Linear Wound Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 902404
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Surgical Wound Cosmesis
Keywords: Cosmesis; Surgical Wound; Fast Absorbing Gut; Linear Cutaneous Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: The primary endpoint will be the score of two blinded reviewers using the patient observer scar assessment score at a three-month assessment visit.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-0 fast absorbing gut suture (Experimental): 6-0 fast absorbing gut used to suture wound
  Interventions: Device: 6-0 fast absorbing gut suture
- 5-0 fast absorbing gut suture (Experimental): 5-0 fast absorbing gut used to suture wound
  Interventions: Device: 5-0 fast absorbing gut suture

INTERVENTIONS:
Device: 6-0 fast absorbing gut suture — Fast absorbing surgical gut suture is a strand of collagenous material, size 6-0
  Arms: 6-0 fast absorbing gut suture
Device: 5-0 fast absorbing gut suture — Fast absorbing surgical gut suture is a strand of collagenous material, size 5-0
  Arms: 5-0 fast absorbing gut suture

SUMMARY:
Traditionally, dermatologic surgeons close wounds with stitches. Fast absorbing gut is a dissolvable stitch that is very commonly used. Some surgeons believe that using a thinner size of this stitch causes less skin reaction and improves the cosmetic outcome of the scar. Other surgeons believe that using a thicker size of this stitch reduces the tension on the scar and improves the cosmetic outcome of the scar in that manner. The investigator wishes to determine whether the thickness of the fast absorbing gut suture that is used makes a difference in the cosmetic outcome of the scar.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the use of 6-0 fast absorbing gut during repair of linear cutaneous surgery wounds on the face or neck improves scar cosmesis compared to wound closure with 5-0 fast absorbing gut. The investigator will use a split wound model, where half of the wound is repaired with 6-0 fast absorbing gut and the other half is repaired with 5-0 fast absorbing gut. Three-months post-surgery, the scar will be measured via the patient observer scar assessment scale, a validated scar instrument. The scar width, and adverse events will also be recorded.

This study aims to investigate whether 5-0 versus 6-0 fast absorbing gut suture leads to better surgical wound cosmesis on the head and neck. The 5-0 fast absorbing gut suture has a large diameter, and therefore greater tensile strength. The greater tensile strength would provide better support of the healing scar during the first 5-7 days after surgery and for this reason, could potentially lead to improved scar cosmesis. However, the greater diameter could also lead to track marks that are larger and more visible. Furthermore, fast absorbing gut has a high degree of tissue reactivity to begin with, and it is known that larger diameter sutures generate more tissue reactivity compared to smaller diameter sutures of the same material; therefore, it is also possible that the 6-0 fast absorbing gut suture would provide better scar cosmesis by virtue of its lower tissue reactivity3,4.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the head and neck with predicted primary closure
* Willing to return for follow up visit.

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Scar Assessment | 3 months following the procedure
  The primary endpoint will be the score of two blinded reviewers using the patient observer scar assessment score at a three-month assessment visit.

SECONDARY OUTCOMES:
Width of the Scar | 3 months following the procedure
  The secondary endpoints will include the width of the scar 1 cm from midline on each side at the follow-up visit and any complications from the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tajirian AL, Goldberg DJ. A review of sutures and other skin closure materials. J Cosmet Laser Ther. 2010 Dec;12(6):296-302. doi: 10.3109/14764172.2010.538413. PMID 21142740
- [Background] Hochberg J, Meyer KM, Marion MD. Suture choice and other methods of skin closure. Surg Clin North Am. 2009 Jun;89(3):627-41. doi: 10.1016/j.suc.2009.03.001. PMID 19465201
- [Background] Gabrielli F, Potenza C, Puddu P, Sera F, Masini C, Abeni D. Suture materials and other factors associated with tissue reactivity, infection, and wound dehiscence among plastic surgery outpatients. Plast Reconstr Surg. 2001 Jan;107(1):38-45. doi: 10.1097/00006534-200101000-00007. PMID 11176599
- [Background] van Rijssel EJ, Brand R, Admiraal C, Smit I, Trimbos JB. Tissue reaction and surgical knots: the effect of suture size, knot configuration, and knot volume. Obstet Gynecol. 1989 Jul;74(1):64-8. PMID 2543937